CLINICAL TRIAL: NCT01100658
Title: Effects of Methylphenidate on Neuropsychological Functioning in Children With Attention Deficits Secondary to Childhood Cancer
Brief Title: Effects of Methylphenidate on Attention Deficits in Childhood Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: University of Minnesota (Other)
Collaborators: Children's Cancer Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2009NTLS075; 0907M69644 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: ALL, Childhood; Leukemia, Lymphoblastic; Leukemia, Lymphoblastic, Acute; Leukemia, Lymphoblastic, Acute, L1; Leukemia, Lymphoblastic, Acute, L2; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive; Leukemia, Lymphocytic, Acute; Leukemia, Lymphocytic, Acute, L1; Leukemia, Lymphocytic, Acute, L2; Lymphoblastic Leukemia; Lymphoblastic Leukemia, Acute; Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Leukemia, Acute, L1; Lymphoblastic Leukemia, Acute, L2; Lymphoblastic Lymphoma; Lymphocytic Leukemia, Acute; Lymphocytic Leukemia, L1; Lymphocytic Leukemia, L2; Brain Tumors; Cancer of the Brain; Cancer of Brain; Malignant Primary Brain Tumors; Brain Neoplasms, Malignant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Brain Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator): Administered 1 capsule each day for 1 week, .3 mg/kg dose.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Administered 1 capsule each day for 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 1 capsule each day for 1 week, .3 mg/kg dose.
  Other Names: Metadae CD (TM); Methylphenidate hydrochloride
  Arms: Methylphenidate
Drug: Placebo — 1 capsule per day for 1 week.
  Other Names: Inactive substance
  Arms: Placebo

SUMMARY:
While neurocognitive impairments in attention, memory and executive functioning are commonly reported sequelae of childhood leukemia and brain tumors, studies have only recently begun to examine the treatment of attention deficits in this population. Numerous studies have examined the effectiveness of methylphenidate in the treatment of children with attention deficit hyperactivity disorder (ADHD). However, the effectiveness of this medication for improving attention and behavioral functioning in children with medical illnesses or brain injury are less clear.

Patients will be randomized to receive one week of Metadate CD (a controlled release form of methylphenidate, similar to Ritalin) and one week of placebo in a double-blind fashion.

ELIGIBILITY:
Inclusion Criteria:

Initial Screening and Registration

* Previous diagnosis of acute lymphoblastic leukemia or brain tumor and have been off treatment and in disease-free remission for a minimum of one year; treated at the University of Minnesota Medical Center, Fairview.
* Proficient in English
* Have given informed consent (assent)

After Initial Screening

* Have evidence of attention impairment based on parent report of attention deficit (> and = 75% on attention deficit hyperactivity disorder [ADHD] Index, Hyperactivity, or Cognitive-Problems/Inattention Index of parent-completed attention deficit hyperactivity disorder (ADHD) rating scale [Conners Parent Rating Scale] and perform at least 1.0 standard deviations below the mean on Omissions, Commissions, or Variability indexes of the Test of Variables of Attention (TOVA)
* Have an estimated Full Scale IQ score on the Wechsler Abbreviated Scale of Intelligence (WASI) >55.

Exclusion Criteria:

* Have optic pathway gliomas and/or neurofibromatosis
* Diagnosed with ADD/ADHD prior to their cancer diagnosis
* Currently taking antidepressants or antipsychotics
* Currently being treated with stimulant medication
* Blind
* Have glaucoma
* Have a family or personal history of motor or phonic tics or Tourette syndrome
* Have seizures not controlled by antiepileptic drugs
* Taking an MAO-inhibitor
* Have a history of cardiovascular disease, uncontrolled hypertension, or hyperthyroidism, or current hypertension requiring antihypertensives

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Kunin-Batson, Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 patient was enrolled in this study. This patient completed baseline assessment, but withdrew from the study before beginning the medication trial. No medications/placebo were administered.
Groups:
- Participant With Attention Deficit: Participant previously had acute lymphoblastic leukemia or brain tumor to be treated with Methylphenidate or Placebo - Administered 1 capsule each day for 1 week, .3 mg/kg dose.
Period: Overall Study
Arm/Group | Participant With Attention Deficit
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participant With Attention Deficit
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Methylphenidate on Neurocognitive Components
Description: Child performance on neuropsychological testing (i.e., using Test of Variables of Attention [TOVA] which is a computerized test of attention that assists in the screening, diagnosis, and treatment monitoring of attention disorders, like Attention Deficit Hyperactivity Disorder [ADHD], and working memory index of the WisSC IV. Standard scores average = 100 +/- 15. Higher scores indicate better performance. Scores < or = 1 SD below the mean represent area of deficit.
Time Frame: Week 1 and Week 2
Population: No patients received treatment, therefore analysis was not done.
Arm/Group | Participant With Attention Deficit
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Parent and Teacher Ratings of Attention, Executive Functioning and Behavior
Description: Parent and teacher ratings of attention, executive function and behavior (i.e., Behavior Rating Inventory of Executive Function [BRIEF -a parent questionnaire and a teacher questionnaire-designed to assess executive functioning in home and school environments. Conners Parent Rating Scale-3 Short Form [CPRS-3 research and clinical tool for obtaining parental reports of childhood behavior problems.] Standard scores average = 50 + or - 10. Higher scores indicate more severe difficulty. Scores > or = 60 represent areas of significant behavior concern.
Time Frame: Week 1 and Week 2
Population: No patients received treatment, therefore analysis was not done.
Arm/Group | Participant With Attention Deficit
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No patients received treatment, therefore no adverse events were reported.
Arm/Group | Participant With Attention Deficit
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Only 1 patient was enrolled in this study, no analysis/outcome data can be reported. This patient completed baseline assessment, but withdrew from the study before beginning the medication trial. No medications/placebo were administered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes